CLINICAL TRIAL: NCT02688257
Title: Assessing Treatment Response of Breast Cancer Using Multimodal Functional Imaging
Brief Title: Assessing Treatment Response in Breast Cancer With Functional Imaging
Status: Completed | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Principal Investigator, NdeSouza, Professor Nandita DeSouza, Institute of Cancer Research, United Kingdom
Other Study IDs: 10/H0806/50 CCR3372
Record Dates: First submitted 2016-02-08; First posted 2016-02-23 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
Keywords: Magnetic Resonance Imaging; Ultrasound; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: MRI — Functional magnetic resonance imaging
Other: Ultrasound — Optoacoustic imaging

SUMMARY:
Patients with large primary operable breast cancers are offered chemotherapy prior to surgery to shrink the tumour and enable breast conserving surgery. Conventional assessment of response to chemotherapy relies on a change in tumour size which does not always correlate with the change in amount of viable tumour. Newer techniques such as functional MRI, microbubble and optoacoustic ultrasound offer the potential to detect responses to chemotherapy by evaluating functional changes in tumour vascularity and oxygenation. Neither modality utilises ionising radiation.

Although MRI is widely used for detecting breast cancer, its ability in assessing functional responses to chemotherapy prior to surgery has not been fully exploited. Dynamic contrast enhanced (DCE) MRI has a sensitivity around 90% and provides quantitative measurements of blood volume and flow. Other functional techniques detect variation in tissue oxygenation: this is called the blood oxygen level-dependent (BOLD) mechanism. The BOLD technique uses a special magnetic resonance (MR) sequence called T2* to measure the weakly magnetic effect of deoxygenated haemoglobin. The investigators wish to develop and validate T2* measurements which relate to oxygenation of a tumour. The investigators also want to validate other MR sequences including diffusion weighted (DW) MRI, which quantifies microcirculation of blood in the capillary network and the diffusion of water within tissues.

Microbubble ultrasound is an established technique that utilises an intravenous contrast agent comprising tiny microbubbles of gas that can increase the reflectivity of blood and enhance spectral and colour Doppler signals obtained from routine ultrasound imaging. Optoacoustic imaging is new technique where the output signal depends on the oxygenation of the tissues under study. It utilises a light signal input and measures ultrasound signal output.

The investigators want to correlate our imaging findings with histopathology after surgical resection of the tumour.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer due for neoadjuvant chemotherapy

Exclusion Criteria:

* Ferromagnetic implants within body in accordance with standard clinical practice
* claustrophobia
* age <18 or >90

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer who are due for neoadjuvant chemotherapy
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Early and late changes of oxygenation and residual cellularity of patients treated with neoadjuvant chemotherapy, measured using the blood oxygen level dependent (BOLD) technique. | 6 years
  The primary aim of the study is to determine whether specific MRI sequences including dynamic contrast enhanced (DCE) MRI, T2*, diffusion weighted (DW) MRI, as well as microbubble and optoacoustic ultrasound imaging provide early measures of treatment response in breast tumours treated with neoadjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Nandita DeSouza, Principal Investigator — ICR
Locations (1):
- The Institute of Cancer Research and Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom